CLINICAL TRIAL: NCT03509610
Title: The Acute Responses to Manipulating Dietary Carbohydrate Content and Type on All Major Aspects of Energy Balance
Brief Title: Acute Responses to Dietary Carbohydrate Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Dr, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP 17/18 87
Record Dates: First submitted 2018-04-09; First posted 2018-04-26 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Nutrition and Energy Balance
Keywords: Nutrition; Carbohydrates
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (Active Comparator): Diet consisting of 50% carbohydrate (20% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOW SUG (Experimental): Diet consisting of 50% carbohydrate (<5% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOW CHO (Experimental): Diet consisting of <8% carbohydrate (<5% sugar), 15% protein, >77% fat
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Macronutrient composition (specifically type and/or amount of carbohydrate) is manipulated

SUMMARY:
Sugar is perceived negatively, leading to government taxation and targets to reduce consumption. These actions have been taken based on the limited evidence that high-sugar diets are associated with greater total energy intake. However, energy intake comprises just one half of the energy balance equation (e.g. balance = intake - expenditure). Without considering energy expenditure, it is impossible to understand the effects of sugar on health. Sugar, and perhaps total carbohydrate intake, may be important for energy balance - perhaps by stimulating increased energy expenditure.

Understanding dietary regulators of energy balance is more important than ever before, because diseases like obesity are a consequence of energy surplus (i.e. energy intake > energy expenditure). No studies have investigated a causal role of dietary sugar or carbohydrate on energy balance. The proposed research will seek to understand the acute (e.g. 24-hour) responses to manipulating dietary carbohydrate and sugar content on energy balance and health.

This research will contribute to enabling individuals to make informed dietary choices about carbohydrate and sugar consumption.

To achieve this, healthy non-obese adults will be recruited to a randomised crossover study. Measures of energy intake, energy expenditure, metabolic health, appetite, food preference, and gut microbiota will be taken. All laboratory trials will take place at the University of Bath.

Three diets will be investigated:

1. Control - reflecting the composition of a typical European diet
2. Low sugar - the same composition of a typical European diet but with <5% energy intake from sugar
3. Low carbohydrate - low carbohydrate diet with <5% energy intake from sugar and <8% energy intake from carbohydrate, replacing carbohydrate energy with fat

The study will consist of a 3-day lead-in period with the control diet followed by one trial day with each diet.

DETAILED DESCRIPTION:
Dietary sugar is increasingly perceived in a negative way. This has led to taxation by government and guidelines by global public health bodies to reduce sugar intake to <5% of energy intake. All available public health guidelines regarding sugar advocate a reduction in sugar intake, despite a lack of evidence to support these recommendations. These guidelines focus on the association between sugar intake and energy intake, without regard for energy expenditure. This oversimplifies situations in which energy surplus is pathological, for example in diseases like obesity. This complexity is demonstrated by evidence that dietary sugar intake is decreasing in the United Kingdom, whilst rates of obesity have increased in the same timeframe.

It is important to consider energy expenditure in the context of health. The most variable component of energy expenditure between individuals is physical activity energy expenditure (PAEE), which varies from ~600-2100 kcal per day in men of a similar demographic. Current guidelines do not regard the effect that changing dietary sugar might have on PAEE and therefore total energy expenditure.

Carbohydrate availability dictates the capacity to perform physical work. However, the role of carbohydrate in regulating physical activity behaviours has only recently been considered. Ingestion of a carbohydrate-rich breakfast causes a significant increase in 24-hour PAEE compared with no breakfast consumption before midday. The magnitude of this difference is greatest prior to midday, near to when carbohydrate had been ingested and when glucose uptake to peripheral tissue is increased. This points towards a stimulatory role of carbohydrate or sugar on PAEE when carbohydrate is readily available to peripheral tissue. The amount of carbohydrate present in skeletal muscle is dictated by the amount of carbohydrate in the diet. As physical activity is performed by skeletal muscle, dietary carbohydrate intake may regulate physical activity behaviour. Consequently, reducing total carbohydrate intake may result in reduced PAEE.

Studies in which carbohydrate has been manipulated and physical activity has been measured have not been sufficient in answering this research question. Often self-report measures of physical activity are used, which are not sensitive enough to discern meaningful differences. Studies which have measured physical activity objectively, i.e. using pedometers or accelerometers, are confounded by a lack of information about actual carbohydrate intake or concurrent prescription of exercise interventions. Furthermore, government targets of reduced sugar intake to <5% of total energy intake are not aimed at overall carbohydrate intake per se. In the breakfast study mentioned, sugar intake was significantly greater amongst individuals who ate breakfast compared with individuals who fasted until midday. Therefore, it is also plausible that a regulatory role of carbohydrate on PAEE may be due to the type of carbohydrate rather than the absolute amount.

If the availability of carbohydrate to peripheral tissue plays a regulatory role on PAEE, then theoretically the effects of manipulating the amount or type of carbohydrate will be detectable acutely, within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-29.9 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase or contraceptive use
* No anticipated changes in diet/physical activity during the study (e.g. holidays or diet plans)

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
24-hour physical activity energy expenditure (kcal/day) | 24 hours
  24-hour physical activity energy expenditure (kcal/day)

SECONDARY OUTCOMES:
24-hour energy intake (kcal/day) | 24 hours
  24-hour energy intake (kcal/day)
Fasting glucose concentrations | 24 hours
  Fasting glucose concentrations in serum samples
Postprandial glucose concentrations | 24 hours
  Postprandial glucose concentrations in serum samples
Fasting insulin concentrations | 24 hours
  Fasting insulin concentrations in serum samples
Postprandial insulin concentrations | 24 hours
  Postprandial insulin concentrations in serum samples
Fasting triglyceride concentrations | 24 hours
  Fasting and postprandial triglyceride concentrations determined in plasma samples
Postprandial triglyceride concentrations | 24 hours
  Postprandial triglyceride concentrations in serum samples
Fasting non-esterified fatty acid concentrations | 24 hours
  Fasting non-esterified fatty acid concentrations in serum samples
Postprandial non-esterified fatty acid concentrations | 24 hours
  Postprandial non-esterified fatty acid concentrations in serum samples
Fasting beta-hydroxybutyrate concentrations | 24 hours
  Fasting beta-hydroxybutyrate concentrations in serum samples
Postprandial beta-hydroxybutyrate concentrations | 24 hours
  Postprandial beta-hydroxybutyrate concentrations in serum samples
Subjective appetite | 24 hours
  Measured by 0-100 mm visual analogue scale
Food preference ratings | 24 hours
  Food preference ratings determined by bespoke computer software
Resting substrate oxidation | 24 hours
  Resting substrate oxidation determined by indirect calorimetry
Postprandial substrate oxidation | 24 hours
  Postprandial substrate oxidation determined by indirect calorimetry
Palatability | 24 hours
  Measured by 0-100 mm visual analogue scale
Fasting cholesterol, HDL, and LDL concentrations | 24 hours
  Fasting cholesterol, HDL, and LDL concentrations in serum samples
Postprandial cholesterol, HDL, and LDL concentrations | 24 hours
  Postprandial cholesterol, HDL, and LDL concentrations in serum samples
Fasting leptin concentrations | 24 hours
  Fasting leptin concentrations in serum samples
Postprandial leptin concentrations | 24 hours
  Postprandial leptin concentrations in serum samples
Macronutrient intake | 24 hours
  Macronutrient intake across 24-h
Fasting FGF21 concentrations | 24 hours
  Fasting FGF21 concentrations in serum samples
Postprandial FGF21 concentrations | 24 hours
  Postprandial FGF21 concentrations in serum samples
Eating rate | 24 hours
  Time taken to eat test meals
Body mass | 24 hours
  Body mass
Waist and hip circumference | 24 hours
  Waist and hip circumference, waist:hip ratio
Fasting haematology profile | 24 hours
  Fasting haematology profile including WBC, RBC, HGB, haematocrit, platelet count

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith HA, Gonzalez JT, Thompson D, Betts JA. Dietary carbohydrates, components of energy balance, and associated health outcomes. Nutr Rev. 2017 Oct 1;75(10):783-797. doi: 10.1093/nutrit/nux045. PMID 29028272
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233
- [Background] Erickson J, Sadeghirad B, Lytvyn L, Slavin J, Johnston BC. The Scientific Basis of Guideline Recommendations on Sugar Intake: A Systematic Review. Ann Intern Med. 2017 Feb 21;166(4):257-267. doi: 10.7326/M16-2020. Epub 2016 Dec 20. PMID 27992898
- [Derived] Hengist A, Davies RG, Rogers PJ, Brunstrom JM, van Loon LJC, Walhin JP, Thompson D, Koumanov F, Betts JA, Gonzalez JT. Restricting sugar or carbohydrate intake does not impact physical activity level or energy intake over 24 h despite changes in substrate use: a randomised crossover study in healthy men and women. Eur J Nutr. 2023 Mar;62(2):921-940. doi: 10.1007/s00394-022-03048-x. Epub 2022 Nov 3. PMID 36326863
- See also: SACN 2015 Report on Carbohydrates and Health — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/445503/SACN_Carbohydrates_and_Health.pdf